CLINICAL TRIAL: NCT05280951
Title: Focused-PPC: An Integrated Postpartum Care, Education, and Support Model for Women in Ghana
Acronym: Focused-PPC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Notre Dame (Other)
Collaborators: Savana Signatures (Unknown); Indiana University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21-06-6662
Record Dates: First submitted 2022-02-10; First posted 2022-03-15 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Postpartum Care
Keywords: postpartum care; postpartum complications; maternal mortality; maternal health; Ghana; postpartum education
MeSH Terms: conditions — Maternal Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Focused-PPC Group (Experimental): Focused-PPC will be implemented in 12 groups (3 groups per health center), with each group having 8 postpartum women. Each group will meet at 1-2 weeks, 6 weeks, and monthly thereafter for up to 1 year postpartum following the Ghana Health Service (GHS) postnatal care schedule.
  Interventions: Other: Focused-PPC Care
- Standard PNC Group (Active Comparator): The control group will contain parallel number of participants as the intervention group in each health center
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Focused-PPC Care — Individual clinical assessments and counseling for each group member will last about 15 minutes. Then, there will be 1 hour of group time dedicated to education and support. Each group session will be led by two trained and registered midwives who will provide both clinical care, education, and support as needed. In addition, each group session will be supported by a project assistant. Focused-PPC will be implemented in addition to newborn care.
  Arms: Focused-PPC Group
Other: Usual Care — Women in the control group will receive standard postnatal care (PNC) currently practiced in the health centers. This involves attending PNC visits at the health center within 14 days after birth, at 6 weeks, and monthly thereafter up to one year.
  Arms: Standard PNC Group

SUMMARY:
The purpose of this project is to test and evaluate an innovative postpartum care, education, and support model that integrates recommended clinical care, education, and support for women in a group setting.

Aim 1. Develop an innovative integrated group postpartum care, education, and support model entitled Focused-PPC for postpartum women up to one year after delivery.

Aim 2. Implement and evaluate this integrated postpartum care model entitled Focused-PPC in a parallel randomized controlled trial with 192 postpartum women at 4 health centers in Tamale, Ghana.

DETAILED DESCRIPTION:
Although the postpartum period poses substantial risks and can result in significant maternal morbidity and mortality, it receives much less attention than pregnancy and childbirth. Appropriate postpartum care enables healthcare providers identify and treat postpartum complications promptly, offer help with a wide range of health and social needs and encourage mothers to adopt evidenced-based postpartum practices at home, since maternal self-care usually takes place at home. In many settings in Sub-Saharan Africa, quality postpartum care, education, and support for the mother are often the missing components of postnatal care delivery, which focuses on care of the baby. The lack of standard postpartum care for the mother contributes to maternal deaths. There is an urgent need for an integrated postpartum care delivery model that is comprehensive and meets clinical care, education, and support needs of mothers. Thus, the purpose of this project is to test and evaluate an innovative postpartum care, education, and support model known as Focused-PPC, in Tamale, Ghana. The proposed project will be the first of its kind to design an integrated and comprehensive group postpartum care delivery model, focused on clinical care of the mother and baby, as well as education and peer support in Ghana. Our model supports the clinical assessments and timeframes recommended by the World Health Organization and adopted by Ghana Health Service. Together with my partner organization, Savana Signatures, we will develop and test Focused-PPC. Focused-PPC will be implemented in groups in health centers in Tamale, Ghana. Each group will meet at 1-2 weeks, 6 weeks, and monthly thereafter for up to 1 year postpartum following the Ghana health service postnatal care schedule. Led by trained midwives in the health centers, each group session will consist of postpartum clinical assessments for mother (in addition to baby), education, and support. Focused-PPC has the potential to change the postpartum care delivery model in Ghana and other countries in sub-Saharan Africa and beyond. Results from this implementation will be used to further refine and scale up the Focused-PPC model of postpartum care.

ELIGIBILITY:
Inclusion Criteria at Recruitment:

* 18 years and older, third trimester of pregnancy, able to understand English or "Dagbani" (the local language)

Inclusion Criteria at Enrollment:

* 18 years and older, had a live birth, able to understand English or "Dagbani" (the local language)

Exclusion Criteria:

* Had a stillbirth

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2022-02-26 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Number of Post-Birth Warning Signs Identified Per Participant | 1 year
  Knowledge of post-birth warning signs will be assessed using a question that asks participants to identify (check all that apply) warning signs of complications. Response options will include nine post-birth warning signs. Each item will be recorded as dichotomous, with a value of 1 assigned if the woman identified the warning sign and 0 if she did not. The total knowledge score will be the sum of these dichotomous items. The mean knowledge score will be calculated as the total knowledge score divided by 9 and reflect the percentage of warning signs known.
  We will model and test the between treatment and control group's knowledge of post-birth warning signs at each timepoint and between timepoints will be assessed using a repeated measure multivariate analysis of variance (MANOVA) with a time and treatment interaction will be run as the primary analysis controlling for baseline demographic variables.

SECONDARY OUTCOMES:
Postpartum Health Behaviors Practiced | 1 year
  Postpartum Health Behaviors will be assessed using a questionnaire. The questionnaire will identify which PNC visits the participant attended, how participants feed their baby, how often the participant adheres to the 4-star diet, feelings on getting pregnant within 6 months of giving birth, plans on getting pregnant within 6 months of giving birth, and intentions on getting pregnant within 6 months of giving birth. The researchers expect health behaviors to be different between the Focused-PPC and control groups. All health behavior questions are all categorical and will be aggregated using latent class analysis.

OTHER OUTCOMES:
postpartum health status | 1 year
  overall health and mental health
Overall Satisfaction of Focused-PPC Sessions | 1 year
  Using a questionnaire, we will record how satisfied participants were with the education received during the Focused-PPC sessions, the clinical care received during the Focused-PPC sessions, whether length of sessions was satisfactory or disliked, whether length of sessions was satisfactory or disliked, whether information provided was satisfactory or disliked, whether peer support was satisfactory or disliked, and whether the group format was liked by participants. These measures are all categorical and will be aggregated using factor analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Yenupini J Adams, PhD, BSN, Principal Investigator — University of Notre Dame
Locations (4):
- Ghana (4):
  - Bagabaga Health Center, Tamale
  - Choggu Health Center, Tamale
  - Kalpohin Health Center, Tamale
  - Kanvilli Health Center, Tamale

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adams YJ, Agbenyo JS, Lau E, Young J, Haas D. Randomized Trial of Group Postpartum Care Model Improves Knowledge and Clinical Outcomes. Nurs Res. 2025 May-Jun 01;74(3):171-178. doi: 10.1097/NNR.0000000000000814. Epub 2025 Feb 13. PMID 39968953
- [Derived] Adams YJ, Agbenyo JS. Improving the Quality of Postpartum Care in Ghana: Protocol for a Parallel Randomized Controlled Trial. JMIR Res Protoc. 2023 Aug 22;12:e47519. doi: 10.2196/47519. PMID 37606965